CLINICAL TRIAL: NCT05968768
Title: To Evaluate the Efficacy and Safety of Naxitamab in Patients With Refractory Ewing's Sarcoma
Brief Title: To Evaluate the Efficacy and Safety of Naxitamab in Patients With Refractory Ewing's Sarcoma (Butterfly)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anna Raciborska (Other)
Collaborators: Wroclaw Medical University (Other)
Responsible Party: Sponsor-Investigator, Anna Raciborska, Prof Ass, Institute of Mother and Child, Warsaw, Poland
Organization: Institute of Mother and Child, Warsaw, Poland (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Butterfly
Record Dates: First submitted 2023-06-13; First posted 2023-08-01 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Ewing Sarcoma
Keywords: Ewing Sarcoma
MeSH Terms: conditions — Sarcoma, Ewing | interventions — naxitamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental - Naxitamab Arm (Experimental): Treatment with naxitamab will be continued no longer than 6 cycles a year or until disease progression, patient consent, unacceptable toxicities, or study closure
  Interventions: Drug: Naxitamab
- Control Group - standard treatment (No Intervention): The control group - will receive only standard treatment.

INTERVENTIONS:
Drug: Naxitamab — Naxitamab will be used only in a hospital setting and must be administered under the supervision of a doctor with experience in the use of oncological therapies. The medicinal product must be administered by a healthcare professional prepared to deal appropriately with severe allergic reactions, including anaphylaxis, in an environment that provides immediate, full access to resuscitation. The patient should have 2 well-functioning IV accesses before any naxitamab treatment is initiated. The solution should be administered through a peripheral or central intravenous catheter. Other concomitant intravenous medicinal products should be administered through separate intravenous access. Before the start of each infusion, premedication will be carried out.
  Other Names: danyelza
  Arms: Experimental - Naxitamab Arm

SUMMARY:
Prospective, interventional, open, randomized, national, multicenter, non-commercial trial

DETAILED DESCRIPTION:
The study includes:

1. Biology screening: to estimate expression on GD2 on Ewing sarcoma cells from tumor tissue from archival material. Availability of tumor tissue is required for pre-screening testing to determine GD2 expression. To be screened for potential enrollment into the study patients or their legal representatives must have signed the pre-screening informed consent form (ICF) to consent to using their archival tumor sample to test the expression of GD2 in their tumor. The expression level of GD2 will be characterized in tumor tissue by immunohistochemistry (IHC) at a local and a central diagnostic testing laboratory.
2. Standard stratifying diagnostic tests (laboratory assessment: morphology, blood chemistry including ALT, AST, eGFR, creatinine, sodium, potassium, coagulation, urine analysis including pH, blood, protein, leukocytes, glucose, urobilinogen, bilirubin, ketones, nitrites, specific gravity, vital signs (body temperature, systolic and diastolic blood pressure, and pulse rate), ECG, cardiac function test, imaging test: CT/MRI scan).
3. Patients with GD2 expression will be randomized in proportions (2:1) to the experimental (D) and control groups (S). The cohort D will consist of 16 subjects, the cohort S 8 subjects. The exploratory cohort D will receive the experimental regimen in 3-week cycles consisting of irinotecan given intravenously (iv) 50 mg/m2 after oral temozolomide 100 mg/m2 on days 1-5 and naxitamab administered iv 2.25 mg/kg/day over 30 - 60 minutes, days 2, 4, 8 and 10 (up to 150 mg/day; total 9 mg/kg per cycle), and GM-CSF 250 mg/m2/day subcutaneously, days 6-10. Patients randomized to arm S will receive IT alone. Treatment cycles will be repeated every 21 days summary to 6 cycles or until disease progression, or subsequent relapsed, or occurrence of intolerable toxicity, or any event making impossible treatment continuation, or investigator's judgment, or withdrawal of consent. All activities are presented in Schedule of Assessments (SoA) at the end of the study synopsis.
4. Patients will be recalculated according to the intent to treat (ITT) rule.
5. The study will be conducted in accordance to GCP and after EC approval of the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven Ewing sarcoma of the bone or soft tissues.
2. Subject's archival tumour sample (formalin-fixed, paraffin-embedded; FFPE) available for evaluation of GD2 expression.
3. Documented disease progression (during or after completion of at least one line treatment) or any subsequent recurrence.
4. GD2 positive tumor assessed by IHC.
5. Age ≥ 2 years and ≤ 21 years.
6. Life expectancy of at least 12 weeks from the time informed consent was signed.
7. Previous systemic anticancer treatment completed ≥ 3 weeks, major surgery ≥ 2 weeks, and radiation therapy ≥ 4 weeks prior to study enrollment.
8. Recovered from adverse effects of prior surgery, radiotherapy, or Clinical trial protocol BUTTERFLY version 1.0 of 30.09.2022 r.anti-neoplastic therapy at the discretion of the investigator.
9. Signing of informed consent for trial participation (including for naxitamab treatment) according with current legal regulations.
10. Consent to the use of effective contraception throughout the period of the study and a minimum of 1 year after discontinuation of study treatment in patients at puberty and sexual maturity

Exclusion Criteria:

1. Failure to meet any of the inclusion criteria.
2. Not eligible to IT.
3. Previous treatment with an anti-GD2 antibody.
4. Hypersensitivity to the study drugs or any of their ingredients (covers IT and naxitamab).
5. Simultaneous treatment with other drugs which might interact with naxitamab or IT regimen.
6. Persistent toxicity related to prior therapy, making it impossible to treat with naxitamab.
7. Significant cardiac conduction abnormalities, including known familial prolonged QT syndrome, or screening corrected QT interval (QTc) >480 msec.
8. Symptoms of congestive heart failure or left ventricular ejection fraction <50%.
9. Inadequate pulmonary function defined as evidence of dyspnea at rest, exercise intolerance, and/or chronic oxygen requirement. In addition, room air pulse oximetry < 94% and/or abnormal pulmonary function tests if these assessments are clinically indicated.
10. Requirement, or likely requirement, for corticosteroids at doses >10 mg prednisolone (or equivalent) per day or other immunosuppressive agents.
11. Diagnosis of other malignancies before study inclusion.
12. Planning to become pregnant (while being treated with IT or naxitamab), pregnancy or breastfeeding.
13. Other acute or persistent disorders, behaviors or abnormal laboratory test results, which might increase the risk related to the participation in this clinical trial or to taking the study drug, or which might influence the interpretation of the study results, or which, in the investigator's opinion, disqualify a patient from participating in the tri

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Safety assessment of the addition of naxitamab to standard 3-week chemotherapy (CHT) in patients with refractory Ewing's sarcoma (ES) | up to 240 days
  Safety will be assessed by number of serious adverse events (SAE), by the number of adverse events (AE), by medical examination with the analysis of recorded vital signs, laboratory abnormalities according to NCI CTCAE v5.0

SECONDARY OUTCOMES:
Event-Free Survival (EFS ) | 3 years
  Will be measured from randomization to death, disease progression or recurrence, or secondary malignancy, whichever comes first
Progression-Free Survival (PFS) | 1 year
  from randomization to progression of the disease
Overall Response Rate (ORR) | 126 days
  Defined as the proportion of patients with a best overall response of complete response (CR) or partial response (PR),
Overall Survival (OS) | 3 years
  Will be measured from randomization to subject's death

CONTACTS AND LOCATIONS:
Overall Officials: Anna Raciborska, Prof., Principal Investigator — the Institue of Mother and Child
Locations (2):
- Poland (2):
  - Mother and Child Institute, Warsaw, Mazowian
  - Wroclaw Medical University, Wroclaw

REFERENCES:
- [Result] Nakajima M, Guo HF, Hoseini SS, Suzuki M, Xu H, Cheung NV. Potent antitumor effect of T cells armed with anti-GD2 bispecific antibody. Pediatr Blood Cancer. 2021 Jul;68(7):e28971. doi: 10.1002/pbc.28971. Epub 2021 Apr 12. PMID 33844437
- [Result] Chan GC, Chan CM. Anti-GD2 Directed Immunotherapy for High-Risk and Metastatic Neuroblastoma. Biomolecules. 2022 Feb 24;12(3):358. doi: 10.3390/biom12030358. PMID 35327550
- [Result] Musumeci F, Cianciusi A, D'Agostino I, Grossi G, Carbone A, Schenone S. Synthetic Heterocyclic Derivatives as Kinase Inhibitors Tested for the Treatment of Neuroblastoma. Molecules. 2021 Nov 23;26(23):7069. doi: 10.3390/molecules26237069. PMID 34885651
- [Result] Wingerter A, El Malki K, Sandhoff R, Seidmann L, Wagner DC, Lehmann N, Vewinger N, Frauenknecht KBM, Sommer CJ, Traub F, Kindler T, Russo A, Otto H, Lollert A, Staatz G, Roth L, Paret C, Faber J. Exploiting Gangliosides for the Therapy of Ewing's Sarcoma and H3K27M-Mutant Diffuse Midline Glioma. Cancers (Basel). 2021 Jan 29;13(3):520. doi: 10.3390/cancers13030520. PMID 33572900
- [Result] Nazha B, Inal C, Owonikoko TK. Disialoganglioside GD2 Expression in Solid Tumors and Role as a Target for Cancer Therapy. Front Oncol. 2020 Jul 7;10:1000. doi: 10.3389/fonc.2020.01000. eCollection 2020. PMID 32733795
- [Result] Hensel J, Metts J, Gupta A, Ladle BH, Pilon-Thomas S, Mullinax J. Adoptive Cellular Therapy for Pediatric Solid Tumors: Beyond Chimeric Antigen Receptor-T Cell Therapy. Cancer J. 2022 Jul-Aug 01;28(4):322-327. doi: 10.1097/PPO.0000000000000603. PMID 35880942
- [Result] Mora J. Autologous Stem-Cell Transplantation for High-Risk Neuroblastoma: Historical and Critical Review. Cancers (Basel). 2022 May 24;14(11):2572. doi: 10.3390/cancers14112572. PMID 35681553